CLINICAL TRIAL: NCT04483362
Title: CanMove: The Feasibility of Implementing a Physical Activity Intervention for Children Undergoing Acute Cancer Treatment
Brief Title: CanMove: A Physical Activity Program for Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: La Trobe University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MurdochCRI
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Pediatric Cancer
Keywords: physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity (Experimental): Behavioural change techniques to promote physical activity
  Interventions: Behavioral: Complex physical activity intervention

INTERVENTIONS:
Behavioral: Complex physical activity intervention — Structured weekly sessions with a Physiotherapist over an 8 week period, including:
  * Evaluation of current levels of physical activity and physical function - including discussion of results
  * Education regarding the importance of physical activity
  * Supervised physical activity session with a physiotherapist
  * Structured weekly sessions applying behavioural change techniques which aim to increase participation in physical activity. Sessions include: provision of activity monitor (Fitbit Inspire), goal setting, monitoring, collaborative problem solving and action plan implementation. Intervention includes additional time allowance of 1 hour per week to assist in implementing action plan items

SUMMARY:
This study will evaluate a physical activity intervention for children during acute cancer treatment. The intervention aims to encourage children to participate in increased levels of physical activity and reduce the amount of time they spend engaged in sedentary activities. This study also aims to evaluate different ways of assessing physical function in order to determine the best outcome measure to use for children during acute cancer treatment.

DETAILED DESCRIPTION:
All participants will receive the intervention which involves weekly sessions with a physiotherapist and the provision of an activity tracker. The sessions will aim to help motivate participants to be more physically active and identify barriers to physical activity in their environment. The activity tracker will be used to set a steps per day goal for the participant to achieve.

The intervention will be assessed for feasibility using aspects of the Bowen Framework. Under this framework the intervention will be evaluated according to different domains:

* Acceptability: To what extent is a new idea, program, process or measure judged as suitable or satisfying
* Demand: To what extent is a new idea, program, process, or measure likely to be used
* Implementation: To what extent can a new program is successfully delivered to intended participants
* Practicality: To what extent can the program can be carried out with intended participants using existing means, resources, and circumstances
* Limited efficiency: Does the a new program show promise of being successful with the intended population

In order to find out the best way to assess physical function, participants will complete 5 different assessments. The results from these assessments will help to determine the best measure to use in this population.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 5-17 years at the time of consent
* Diagnosed (or relapsed) with cancer >4 weeks and <6 months at time of consent
* Currently receiving cancer treatment at the Royal Children's Hospital
* Has been an in-patient for >7 consecutive days at the time of consent
* Provide a signed and dated informed consent form and/or has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf

Exclusion Criteria:

* Deemed by the treating medical team as unsafe to participate
* Child/adolescent unable to mobilise independent of clinical staff assistance, as classified by the research team at the time of consent (use of a gait aid or assistance from a primary carer/support person is accepted). For example, if a child/adolescent requires assistance from nursing staff or physiotherapist in order to walk, they will be excluded.
* Child/adolescent unable to follow simple instructions
* Suitable support person (18 years and over) not available to participate in continuous monitoring of daily steps in tandem with the child/adolescent
* No suitable access to a device to sync with a Fitbit
* Inability or unwillingness of participant or legally acceptable representative to give written informed consent.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Demand for the intervention | Through completion of recruitment, estimated as 9 months
  Recruitment rate (comparing the number of people recruited to the number of potentially eligible participants), and documenting the reasons for non-participation.
Acceptability of the intervention according to participants | After completion of the intervention (on average 8 weeks)
  Participant and participant guardian perspective on intervention satisfaction and potential areas of improvement via semi-structured interviews
Acceptability of the intervention according to staff | Through study completion, estimated as 1 year
  Staff perspective on intervention satisfaction and potential areas of improvement via focus groups with staff members
Implementation of the intervention: adherence to wearing Fitbit | Post intervention (on average 8 weeks)
  Adherence to wearing the Fitbit for monitoring, percentage of complete Fitbit data days out of total intervention days
Implementation of the intervention: attendance to intervention sessions | Post intervention (on average 8 weeks)
  Adherence to attending intervention sessions, percentage of intervention sessions that were attended
Implementation of the intervention: ability for participants to attain their steps per day goal | Post intervention (on average 8 weeks)
  Goal attainment, percentage of days out of total intervention days that participant was able to achieve their steps per day target
Practicality of the intervention: adverse events | Post the participant's final trial visit (on average 12 weeks)
  Measured by number of adverse events reported related to trial procedures. At each trial visit, participants will be asked "How have you felt since your last visit?" in order to elicit any changes in their well-being. They will also be asked if they have had any falls, new injuries, felt distress as a result of the intervention or experienced a change in medical or mobility status. Adverse events relevant to participant safety will also be documented from correspondence from their primary care physician or from the medical record. Adverse events recorded as serious or non-serious, related or not related to the intervention.
Limited efficiency testing assessing changes in physical activity between pre and post intervention: Actigraph steps per day | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in average steps taken per day measured via the Actigraph
Limited efficiency testing assessing changes in physical activity between pre and post intervention: Fitbit steps per day | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in average steps taken per day measured via the Fitbit
Limited efficiency testing assessing changes in physical activity between pre and post intervention: Actigraph distance travelled per day | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in average distance travelled per day measured via the Actigraph
Limited efficiency testing assessing changes in physical activity between pre and post intervention: Fitbit distance travelled per day | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in average distance travelled per day measured via the Fitbit
Limited efficiency testing assessing changes in physical activity between pre and post intervention: Actigraph physical activity intensity | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in time spent in different physical activity intensities (sedentary, light, moderate-vigorous and vigorous) measured by the Actigraph
Limited efficiency testing assessing changes in physical activity between pre and post intervention: Fitbit physical activity intensity | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in time spent in different physical activity intensities (sedentary, light, moderate-vigorous and vigorous) measured by the Fitbit
Limited efficiency testing assessing changes in physical activity between pre and post intervention: sedentary bouts | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in number of sedentary bouts per day measured via the Actigraph
Limited efficiency testing assessing changes in physical activity between pre and post intervention: body position | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in time spent in each body position per day measured via the Actigraph
Limited efficiency testing assessing changes in physical activity between pre and post intervention: active hours | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in number of active hours per day measured via the Fitbit
Limited efficiency testing assessing changes in physical activity between pre and post intervention: active minutes | Post intervention (on average 8 weeks)
  Mean change from pre to post intervention in number of active minutes per day measured via the Fitbit

SECONDARY OUTCOMES:
Limited efficiency testing assessing changes in physical function from pre to post intervention: Movement ABC | Post intervention (on average 8 weeks)
  Mean score and percentile ranking measured via on the Movement ABC (a performance measure of physical function)
Limited efficiency testing assessing changes in physical function from pre to post intervention: 6 Minute Walk Test | Post intervention (on average 8 weeks)
  Mean distance travelled measured via on the 6 Minute Walk test (a performance measure of physical fitness)
Limited efficiency testing assessing changes in physical function from pre to post intervention: Timed Up and Go | Post intervention (on average 8 weeks)
  Mean time measured via the Timed Up and Go (a performance measure of physical function)
Limited efficiency testing assessing changes in physical function from pre to post intervention: Timed Up and Down Stairs | Post intervention (on average 8 weeks)
  Mean time measured via the Timed Up and Down Stairs (a performance measure of physical function)
Limited efficiency testing assessing changes in physical function from pre to post intervention: Time to Rise from the Floor | Post intervention (on average 8 weeks)
  Mean time and rating for quality of movement measured via the 30 second Chair Stand Test Assessment (a performance measure of physical function)
Limited efficiency testing assessing changes in physical function from pre to post intervention: Time to Rise from the Floor | Post intervention (on average 8 weeks)
  Mean time and rating for quality of movement measured via the Time to Rise from the Floor Assessment (a performance measure of physical function)
Limited efficiency testing assessing changes in Health-related Quality of Life from pre to post intervention: self-reported Pediatric Quality of Life Inventory-core generic module | Post intervention (on average 8 weeks)
  Mean score recorded on the self-reported Pediatric Quality of Life Inventory-core generic module (standardised questionnaire). Items are scored on a 0-100 scale, so that higher scores indicate better health-related quality of life
Limited efficiency testing assessing changes in Health-related Quality of Life from pre to post intervention: proxy-reported Pediatric Quality of Life Inventory-core generic module | Post intervention (on average 8 weeks)
  Mean score recorded on the proxy-reported Pediatric Quality of Life Inventory-core generic module (standardised questionnaire). Items are scored on a 0-100 scale, so that higher scores indicate better health-related quality of life
Feasibility: Limited efficiency testing assessing changes in Health-related Quality of Life from pre to post intervention: self-reported PedsQL-cancer module | Post intervention (on average 8 weeks)
  Mean score recorded on the self-reported Pediatric Quality of Life Inventory-cancer module (standardised questionnaire). Items are scored on a 0-100 scale, so that higher scores indicate better health-related quality of life
Feasibility: Limited efficiency testing assessing changes in Health-related Quality of Life from pre to post intervention: proxy-reported PedsQL-cancer module | Post intervention (on average 8 weeks)
  Mean score recorded on the proxy-reported Pediatric Quality of Life Inventory-cancer module (standardised questionnaire). Items are scored on a 0-100 scale, so that higher scores indicate better health-related quality of life
Categorisation and frequency of reported barriers to physical activity | Post intervention (on average 8 weeks)
  Categorise and collate the frequency of participant reported barriers to physical activity. Data collected during each week of the intervention period
Categorisation and frequency of action plan strategies | Post intervention (on average 8 weeks)
  Categorise and collate the frequency of action plan items put in place to overcome barriers to physical activity. Data collected during each week of the intervention period
Utility of physical function assessment tools, measured by completeness of assessment data for physical function | Post completion of follow up assessment (on average 10 weeks)
  The percentage of physical function assessments that were completed
Utility of physical activity assessment tools, measured by completeness of assessment data for physical activity | Post completion of follow up assessment (on average 10 weeks)
  Percentage of complete Fitbit and Actigraph data days out of total assessment days

OTHER OUTCOMES:
Construct validity of physical function measures | Post completion of follow up assessment (on average 10 weeks)
  Correlation between scores of all physical function measures: Timed up and Go, Movement ABC, Timed Up and Down Stairs, 6 Minute Walk Test, Time to Rise from the Floor
Interpretability of physical function measures | Post completion of follow up assessment (on average 10 weeks)
  Interpretability assessment of all physical function measures used in the trial: Timed up and Go, Movement ABC, Timed Up and Down Stairs, 6 Minute Walk Test, Time to Rise from the Floor
Responsiveness of physical function measures | Post completion of follow up assessment (on average 10 weeks)
  Correlation in mean change over two time points between all physical function measures used in the trial: Timed up and Go, Movement ABC, Timed Up and Down Stairs, 6 Minute Walk Test, Time to Rise from the Floor and Global Rating of Change Score
Criterion validity of physical activity measured on the Fitbit and Actigraph | Post completion of follow up assessment (on average 10 weeks)
  Correlation of physical activity data between Fitbit and Actigraph

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Grimshaw, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital, Parkville, Victora, Australia

IPD SHARING:
Plan to Share IPD: Yes
The participants will be asked to voluntarily consent to data sharing. Beginning from 3 months after article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access:
  * Individual de-identified participant data that underlie the results reported in this article (text, tables, figures and appendices)
  * Trial protocol, Statistical Analysis Plan, Participant Informed Consent Form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months following publication - until the end of archival period (15 year post-trial completion (TGA) or until child aged 25 years (whichever is the later))
Access Criteria: Research projects that have been approved by a Human Research Ethics Committee

REFERENCES:
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699